CLINICAL TRIAL: NCT01848054
Title: A Randomized, Blinded, Active-controlled Non-inferiority Study of the Efficacy and Safety of OX219 for the Induction of Treatment of Opioid Dependence
Brief Title: Study to Assess Efficacy and Safety of BNX Sublingual Tablets for the Induction of Treatment of Opioid Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orexo AB (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OX219-007
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Results first posted 2015-06-24 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Opioid-Related Disorders; Opiate Dependence
Keywords: opioid dependence, buprenorphine/naloxone, sublingual
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BNX Sublingual Tablets Induction (Experimental): Day 1-2 (Blinded Induction): BNX sublingual tablets
  Day 3-28 (Open-label Maintenance): BNX sublingual tablets
  Interventions: Drug: Buprenorphine/naloxone sublingual tablets
- Buprenorphine Induction (Active Comparator): Day 1-2 (Blinded Induction): Generic buprenorphine sublingual tablets
  Day 3-28 (Open-label Maintenance): BNX sublingual tablets
  Interventions: Drug: Buprenorphine/naloxone sublingual tablets; Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine/naloxone sublingual tablets — Advanced-formulation buprenorphine/naloxone sublingual tablets
  Other Names: Zubsolv; OX219
Drug: Buprenorphine — Buprenorphine sublingual tablets
  Other Names: Generic buprenorphine
  Arms: Buprenorphine Induction

SUMMARY:
The purpose of the study was to assess the efficacy of induction treatment with buprenorphine/naloxone (BNX) sublingual tablet s compared with induction treatment with buprenorphine only. The hypothesis is that starting directly on OX219 works equally well (e.g. not significantly worse) as starting on buprenorphine only and switching to OX219 on Day 3.

DETAILED DESCRIPTION:
This was a prospective, randomized, multicenter, blinded, parallel-group, active-controlled, non-inferiority study conducted at 13 sites within the US. Eligible patients participated in 8 treatment visits on Days 1, 2, 3, 4, 8, 15, 22, and 29. Effectiveness of treatment was assessed as follows:

* Retention in treatment at Day 3
* Clinician and patient assessments of opioid withdrawal symptoms
* Assessment opioid cravings

ELIGIBILITY:
Inclusion Criteria:

* Able to read, comprehend, and sign the informed consent form and willingly provide written informed consent
* Prepared to engage in opioid replacement therapy and to abstain from opioid utilization other than the study drug, and from other illicit drugs
* Male or female, 18 to 65 years of age (inclusive)
* Met clinical criteria for opioid dependence in past 12 months based on DSM-IV-TR
* Provided buprenorphine-negative urine drug screen prior to randomization
* Provided negative urine pregnancy test
* Females of childbearing potential were required to be using a reliable method of contraception (e.g., hormonal, condom with spermicide, intrauterine device [IUD]) after the screening visit and for the duration of the study
* Participants receiving opioids for pain must receive clearance from their prescribing physician to be withdrawn from their prescribed opioids
* Generally good health as determined by the investigator
* Participants should demonstrate at least mild withdrawal symptoms (defined as a COWS score >9 at Day 1 predose)

Exclusion Criteria:

* Females who are pregnant or lactating, or planning to be pregnant during study
* Any previous prescribed treatment with buprenorphine monotherapy (e.g., generic buprenorphine sublingual tablets)
* Prescribed treatment with buprenorphine or naloxone within 90 days prior to start of treatment
* Methadone patients with any daily dose over 30 mg during the past week and who received the last dose of methadone less than 30 hours prior to start of treatment
* Participants who are unwilling or unable to comply with the requirements of the protocol
* Participants who are participating in any other clinical study in which medication(s) are being delivered or who have used an investigational drug or device within the last 30 days
* Participants with any known allergy or sensitivity or intolerance to buprenorphine, naloxone, or any related drug
* Participants who are on the staff, affiliated with, or a family member of the staff personnel directly involved with this study
* Participants with serious untreated Axis I DSM-IV-TR psychiatric comorbidity
* Tongue piercing or other piercings in the mouth, including lips and cheek
* Participants with current or history of clinically significant medical disorder or condition
* Participants who are human immunodeficiency virus (HIV)-seropositive with a CD4+ count <200 or active acquired immune deficiency syndrome (AIDS)
* Participants who have any Class III or IV congestive heart failure, symptomatic myocardial ischemia, a history of long QT syndrome.
* Participants who are currently taking Class 1A antiarrhythmic medications or Class III antiarrhythmic medications
* Participants who have uncontrolled hypertension or clinically significant ECG abnormalities
* Participants who have a pulse oximetry ≤93% at screening, due to any medical reason.
* Individuals with AST or ALT levels ≥3 X the upper limit of normal or total bilirubin or creatinine ≥1.5 X ULN, on the screening laboratory assessments
* Participants with known significant liver disease.
* Participants who take any medication, nutraceutical, herbal product with known CYP3A4 inhibition or induction properties within 14 days of screening.
* Participants who are at suicidal risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Webster, Principal Investigator — Life Tree Pain Clinic, 3838 S 700 E Suite 200, Salt Lake City, UT 84106
Locations (14):
- United States (14):
  - Birmingham, Alabama
  - Haleyville, Alabama
  - National City, California
  - Oceanside, California
  - Jacksonville, Florida
  - Maitland, Florida
  - North Miami, Florida
  - Baltimore, Maryland
  - Fall River, Massachusetts
  - Flowood, Mississippi
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 313 patients were enrolled. Three patients who were randomized did not receive study drug, making the participant flow 310.
Groups:
- BNX Sublingual Tablets Induction: Days 1-2: Induction on BNX sublingual tablets (blinded); Days 3-28: Maintenance treatment with BNX sublingual tablets (open-label)
- Buprenorphine Induction: Days 1-2: Induction on buprenorphine sublingual tablets (blinded); Days 3-28: Maintenance treatment with BNX sublingual tablets (open-label)
Period: Induction Phase
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction
Started | 155 | 155
Completed | 132 | 147
Not Completed | 23 | 8
Period: Stabilization/Maintenance
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction
Started | 132 | 147
Completed | 92 | 107
Not Completed | 40 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction | Total
Number analyzed (Participants) | 155 | 155 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (10.6) | 38.0 (10.9) | 38.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 52 | 107
  Male | 100 | 103 | 203
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 19 | 38
  White | 134 | 135 | 269
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (6.7) | 25.3 (5.0) | 25.7 (5.9)
Duration of opioid dependence [Mean (Standard Deviation); unit: years] | 13.3 (9.3) | 11.6 (9.2) | 12.4 (9.3)

OUTCOME MEASURES:

1. Primary Outcome: Retention in Treatment in the Per Protocol Population
Description: Retention in treatment at Day 3 in the per protocol population (n=256) was defined as the number of patients in each induction arm completing the induction phase and who received study medication on Day 3. Treatment with BNX sublingual tablets was considered non-inferior to generic buprenorphine if the lower limit of the 95% confidence interval for the difference between BNX and generic buprenorphine was ≥-10% in the number of patients retained in treatment on Day 3.
Time Frame: Day 3
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction
Number analyzed (Participants) | 128 | 128
participants | 113 | 122
Statistical Analysis 1: Comparison: BNX Sublingual Tablets Induction vs Buprenorphine Induction; Test type: Non-Inferiority or Equivalence — The primary efficacy analysis of retention in treatment at Day 3 was assessed in the per protocol population. In addition, a sensitivity analysis assessed retention in treatment in the full analysis population. For these assessments, the margin to determine non-inferiority (i.e., lower limit of the 95% CI for the difference between BNX and generic buprenorphine of ≥-10%) was selected based on clinical experience to justify comparison between the 2 treatments; p < 0.05, t-test, 2 sided; Comparisons between treatment groups were reported with 2-sided p values using 95% CIs for the difference

2. Secondary Outcome: Area Under the Curve (AUC) in Clinical Opiate Withdrawal Scale (COWS) Total Score on Days 1 to 3 Inclusive
Description: Least squares mean AUC in COWS total score on Days 1 to 3; COWS scores range from 0-48, with a lower score being more favorable
Time Frame: Pre-dose on Days 1-3 and 0.5, 1, 1.5, 3, and 6 hours post-dose on Day 1
Population: Full analysis population
Measure: Least Squares Mean (Standard Deviation); unit: score x hour
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction
Number analyzed (Participants) | 154 | 154
score x hour | 7.21 (4.3) | 6.88 (4.0)

3. Secondary Outcome: AUC in Subjective Opiate Withdrawal Scale (SOWS) Total Score on Days 1 to 3 Inclusive
Description: Least squares mean AUC day 1 pre-dose through Day 3 in SOWS; SOWS scores range from 0-64, with a lower score being more favorable
Time Frame: Pre-dose on Days 1-3 and 0.5, 1, 1.5, 3, and 6 hours post-dose on Day 1
Population: Full analysis population; patients with missing data were excluded from the analysis and are reflected in the number of participants analyzed
Measure: Least Squares Mean (Standard Deviation); unit: score x hour
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction
Number analyzed (Participants) | 147 | 153
score x hour | 17.7 (13.5) | 17.4 (12.8)

4. Secondary Outcome: AUC in Visual Analog Scale (VAS) Score for Craving on Days 1 to 3 Inclusive
Description: Least squares mean AUC measurement in VAS score for cravings on Days 1 to 3; the VAS craving scores range from 0 ("no cravings") to 100 ("most intense craving I have ever had")
Time Frame: Pre-dose on Days 1-3 and 0.5, 1, 1.5, 3, and 6 hours post-dose on Day 1
Population: as for outcome 3
Measure: Least Squares Mean (Standard Deviation); unit: score x hour
Groups:
- Buprenorphine Induction: Days 1-2: Induction on buprenorphine sublingual tablets (blinded); Days 3-28: Maintenance treatment with OX219 buprenorphine/naloxone sublingual tablets (open-label)
  OX219 buprenorphine/naloxone: OX219 buprenorphine/naloxone sublingual tablets
  Buprenorphine: Buprenorphine sublingual tablets
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction
Number analyzed (Participants) | 153 | 155
score x hour | 40.0 (25.3) | 39.5 (24.7)

5. Secondary Outcome: Mean Change From Baseline in COWS Total Score After Day 3 (Maintenance Phase)
Description: Mean change from baseline in COWS total scores during the maintenance phase (Days 4, 8, 15, 22, and 29); COWS scores range from 0-48, with a lower score being more favorable
Time Frame: Predose on Days 4, 8, 15, 22, and 29
Population: Full analysis population; patients with missing data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- BNX Sublingual Tablets Induction: Days 1-2: Induction on BNX sublingual tablets (blinded); Day 3-28: Maintenance treatment with BNX sublingual tablets (open-label)
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction
Number analyzed (Participants) | 155 | 155
units on a scale
  Day 4 | -9.4 (5.8) | -8.5 (5.7)
  Day 8 | -11.2 (4.9) | -10.1 (5.3)
  Day 15 | -11.9 (4.9) | -11.1 (5.2)
  Day 22 | -12.5 (4.7) | -11.6 (5.0)
  Day 29/premature discontinuation | -12.5 (5.2) | -11.4 (5.4)

6. Secondary Outcome: Mean Change From Baseline in SOWS Total Score After Day 3 (Maintenance Phase)
Description: Mean change from baseline in SOWS total scores during the maintenance phase (Days 4, 8, 15, 22, and 29); SOWS scores range from 0-64, with a lower score being more favorable
Time Frame: Pre-dose on Days 4, 8, 15, 22, and 29
Population: Full analysis population; patients with missing data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- BNX Induction: Days 1-2: Induction on BNX sublingual tablets (blinded); Days 3-28: Maintenance treatment with BNX sublingual tablets (open-label)
Arm/Group | BNX Induction | Buprenorphine Induction
Number analyzed (Participants) | 155 | 155
units on a scale
  Day 4 | -24.7 (16.0) | -18.9 (13.8)
  Day 8 | -27.0 (15.8) | -21.3 (13.6)
  Day 15 | -29.2 (15.5) | -23.3 (13.7)
  Day 22 | -30.8 (15.6) | -24.1 (13.8)
  Day 29/premature discontinuation | -30.4 (16.0) | -24.3 (14.2)

7. Secondary Outcome: Mean Change From Baseline in the VAS Score for Cravings After Day 3 (Maintenance Phase)
Description: Mean change from baseline in VAS scores for cravings during the maintenance phase (Days 4, 8, 15, 22, and 29); the VAS craving scores range from 0 ("no cravings") to 100 ("most intense craving I have ever had")
Time Frame: Pre-dose on Days 4, 8, 15, 22, and 29
Population: Full analysis population; patients with missing data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction
Number analyzed (Participants) | 155 | 155
units on a scale
  Day 4 | -40.1 (28.6) | -34.2 (29.4)
  Day 8 | -46.1 (29.5) | -39.9 (27.7)
  Day 15 | -48.5 (30.3) | -44.3 (26.1)
  Day 22 | -53.3 (29.5) | -47.2 (25.3)
  Day 29 | -52.7 (29.1) | -45.1 (29.8)

8. Secondary Outcome: Retention in Treatment in the Full Analysis Population
Description: Retention in treatment at Day 3 in the full analysis population (N=310) was defined as the number of patients in each induction arm completing the induction phase and who received study medication on Day 3. Treatment with BNX sublingual tablets was considered non-inferior to generic buprenorphine if the lower limit of the 95% confidence interval for the difference between BNX and generic buprenorphine was ≥-10% in the number of patients retained in treatment on Day 3.
Time Frame: Day 3
Population: Full analysis population; patients with missing data were excluded from the analysis
Measure: Number; unit: participants
Groups:
- Buprenorphine Induction: Days 1-2: Induction on buprenorphine sublingual tablets (blinded); Days 3-28: Maintenance treatment with OX219 buprenorphine/naloxone sublingual tablets (open-label)
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction
Number analyzed (Participants) | 155 | 155
participants | 132 | 147
Statistical Analysis 1: Comparison: BNX Sublingual Tablets Induction vs Buprenorphine Induction; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, t-test, 2 sided; Comparisons between treatment groups were reported with 2-sided p values using 95% CIs for the difference

ADVERSE EVENTS:
Time Frame: Blinded Induction Phase (Days 1-2) and Open Label Maintenance Phase (Days 3-28)
Description: The safety population included 310 patients.
Arm/Group | BNX Sublingual Tablets Induction | Buprenorphine Induction
Serious Adverse Events (participants affected / at risk) | 1/155 | 2/155
Other Adverse Events (participants affected / at risk) | 37/155 | 43/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNX Sublingual Tablets Induction (N=155) | Buprenorphine Induction (N=155)
Diabetic ketoacidosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Considered unrelated to study treatment; reported during the blinded induction phase
Attempted suicide (Psychiatric disorders) | 0 (0) | 1 (1) — Considered unrelated to study treatment; reported during the open-label maintenance phase
Bacteremia secondary to pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) — Considered unrelated to study treatment; reported during the open-label maintenance phase
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNX Sublingual Tablets Induction (N=155) | Buprenorphine Induction (N=155)
Nausea (Induction) (Gastrointestinal disorders) | 12 (12) | 13 (13) — Adverse events reported during the blinded induction phase
Headache (Induction) (Nervous system disorders) | 11 (11) | 11 (11) — Adverse events reported during the blinded induction phase
Insomnia (Induction) (Psychiatric disorders) | 6 (6) | 11 (11) — Adverse events reported during the blinded induction phase
Vomiting (Induction) (Gastrointestinal disorders) | 8 (8) | 8 (8) — Adverse events reported during the blinded induction phase

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No